CLINICAL TRIAL: NCT06879613
Title: Comparing Breastmilk, Massage, and no Intervention for Pain Management During Vaccination of Term Infants at the Bamenda Regional Hospital
Brief Title: Comparing Breastmilk, Massage, and no Intervention for Pain Management During Vaccination of Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bamenda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/0030H/UBa/IRB
Record Dates: First submitted 2024-12-06; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breastmilk arm (Experimental): Breastmilk was administered for pain
  Interventions: Dietary Supplement: Breastmilk
- Massage arm (Experimental): Massage was administered for pain
  Interventions: Procedure: Massage
- No interention arm (No Intervention): No intervention was done for pain

INTERVENTIONS:
Dietary Supplement: Breastmilk — Breastmilk from the mother of the infant was given for pain
  Arms: Breastmilk arm
Procedure: Massage — The spot that was vaccinated was massaged by the mother/carer of the infant
  Arms: Massage arm

SUMMARY:
The goal of this clinical trial is to learn if breastmilk, massage or no intervention works for pain management during vaccination of term infants. It will also learn about the safety of these 3 approaches. The main questions it aims to answer is:

Does breastmilk, massage or no intervention works for pain management during vaccination of term infants?

Researchers will compare breastmilk, massage or no intervention for pain management during vaccination of term infants.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at or after 37 completed weeks of gestation.
* Neonates scheduled to receive the DTC-HepB-Hib-1 immunization.
* Time from last feeding should be greater than or equal to 30 minutes.

Exclusion Criteria:

* Term neonates with major congenital abnormalities like limb contractures, limb deformities.
* Term neonates with any neurological conditions like hydrocephalus, cerebral palsy or birth asphyxia.
* Infants with acute illness.
* Infants randomized for no intervention but mothers breastfeed before pain evaluation to calm the babies from crying.

Ages: 6 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Neonatal infant pain score (NIPS) | The pain scores for all the arms was done 2 minutes before vaccination and 30 seconds after vaccination
  The pain score assessment based on the neonatal infant pain score (NIPS). Interpretation: minimum score of 0 and a maximum score of 7. 0-1: no pain; 2: mild pain; 3-4: moderate pain; 5-7: severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Bamenda Regional Hospital, Bamenda, Northwest Region, Cameroon